CLINICAL TRIAL: NCT06272123
Title: Comparison of Endotypic Stability in Various Populations With Chronic Sinusitis
Brief Title: Endotypic Stability in CRS
Status: Recruiting | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 20D.776
Record Dates: First submitted 2024-01-23; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Chronic Sinusitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Sinusitis
  Interventions: Other: no intervention
- Controls
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
A Case control study with 150 cases and 50 controls will be conducted. Immunologic (cytokines measurements in nasal secretions and sinonasal tissues), histopathologic (tissue eosinophilia) and clinical parameters (Lund-Mackay and Lund-Kennedy score, lung function tests), surveys (SNOT- 22, SF-36 quality of life survey) will be compared between different groups of patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic sinusitis (with or without polyps)
* Undergoing endoscopic sinus surgery during the study period
* More than 18 years
* No chronic illness/ malignancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic sinusitis (with or without polyps) undergoing endoscopic sinus surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Endotypic markers | 1 year
  The primary outcome measure assessed through this study is the presence of endotypic markers including: IL-5, IFN-gamma, IL-17a, TNF-alpha, and IL-22 in tissue biopsy samples across multiple racial/ethnic groups.

SECONDARY OUTCOMES:
SF-36 | 1 year
  Differences in SF-36 scores between ethnic groups.
SNOT-22 | 1 year
  Differences in SNOT-22 scores between ethnic groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Department of Otolaryngology, Philadelphia, Pennsylvania, United States